CLINICAL TRIAL: NCT01121146
Title: A Prospective, Randomized Clinical Study Comparing Marathon Polyethylene and Enduron Polyethylene Acetabular Liners Used in Total Hip Arthroplasty
Brief Title: Study Comparing Marathon Polyethylene and Enduron Polyethylene Acetabular Liners Used in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, C. Anderson Engh, Jr., MD, Investigator, Anderson Orthopaedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AORI2010-0100
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
Keywords: Osteolysis; Polyethylene; Crosslinked Polyethylene; Total Hip Replacement; CT
MeSH Terms: conditions — Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Osteolysis | interventions — Arthroplasty, Replacement, Hip

ARMS (2):
- Crosslinked Marathon polyethylene (Active Comparator)
  Interventions: Device: Total Hip Replacement
- Standard Enduron polyethylene (Active Comparator)
  Interventions: Device: Total Hip Replacement

INTERVENTIONS:
Device: Total Hip Replacement — Comparison of Marathon and Enduron polyethylene

SUMMARY:
The purpose of the study is to determine whether crosslinked Marathon and standard Enduron polyethylene liners show differences in bone loss around the hip implant.

DETAILED DESCRIPTION:
Several institutions report very low wear rates with highly crosslinked polyethylene based on early clinical data. However, since bone loss typically appears after 5-year follow-up, the reduction in the incidence and extent of bone loss among total hip replacement patients with crosslinked Marathon liners, compared to those with standard Enduron liners, has not been as dramatic as the wear reduction. Despite the substantial reduction in wear that we observed at 5-year follow-up, the patients' perceptions of their outcomes remained similar among the Marathon and Enduron groups. This study will evaluate outcome at a minimum of 10-years after surgery among the same group of patients whose outcome was previously reported at 5-year follow-up. At 10-year follow-up, we anticipate that the reduction in wear associated with Marathon polyethylene will be associated with significant reductions in bone loss when compared to the Enduron polyethylene.

ELIGIBILITY:
Inclusion Criteria:

(from original study)

-Elective total hip replacement patient

(from 10-year follow-up)

* Consented to the original study.
* Received a Duraloc 100 cup with either a crosslinked Marathon or standard Enduron liner.
* Received an AML/Solution or a Prodigy stem with 28mm cobalt chrome femoral head.

Exclusion Criteria:

(from original study)

-None

(from 10-year follow-up)

* Patient did not receive device as specified in inclusion criteria.
* Patient refused to consent to the 10-year follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 1998-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles A. Engh, Sr., MD, Principal Investigator — Anderson Orthopaedic Research Institute; C. Anderson Engh, Jr., MD, Principal Investigator — Anderson Orthopaedic Research Institute
Locations (1):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States

REFERENCES:
- [Result] Leung SB, Egawa H, Stepniewski A, Beykirch S, Engh CA Jr, Engh CA Sr. Incidence and volume of pelvic osteolysis at early follow-up with highly cross-linked and noncross-linked polyethylene. J Arthroplasty. 2007 Sep;22(6 Suppl 2):134-9. doi: 10.1016/j.arth.2007.04.006. Epub 2007 Jul 27. PMID 17823032
- [Result] Engh CA Jr, Stepniewski AS, Ginn SD, Beykirch SE, Sychterz-Terefenko CJ, Hopper RH Jr, Engh CA. A randomized prospective evaluation of outcomes after total hip arthroplasty using cross-linked marathon and non-cross-linked Enduron polyethylene liners. J Arthroplasty. 2006 Sep;21(6 Suppl 2):17-25. doi: 10.1016/j.arth.2006.05.002. PMID 16950057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Starting in January 1999 for a period of 18 months, patients were enrolled from an orthopaedic clinic.
Pre-assignment Details: Six subjects (6 hips) who had consented to participate were excluded from the study at the time of surgery because they did not receive a hip implant consisting of a 28-mm femoral head and a Duraloc 100 cup with a 4-mm lateralized liner due to intra-operative hip stability, leg length or cup fixation issues.
Groups:
- Crosslinked Marathon Polyethylene: Implanted with a metal femoral head and a crosslinked polyethylene liner.
- Standard Enduron Polyethylene: Implanted with a metal femoral head and a non-crosslinked polyethylene liner.
Period: Overall Study
Arm/Group | Crosslinked Marathon Polyethylene | Standard Enduron Polyethylene
Started | 116 | 114
Completed | 90 (The 90 hips include those that were not revised and had a minimum 9-year questionnaire or radiograph) | 72 (The 72 hips include those that were not revised and had a minimum 9-year questionnaire or radiograph)
Not Completed | 26 | 42
Not completed — Death | 17 | 15
Not completed — Adverse Event | 2 | 11
Not completed — Lost to Follow-up | 7 | 16

BASELINE CHARACTERISTICS:
Groups:
- Crosslinked Marathon Polyethylene; Standard Enduron Polyethylene: Total Hip Replacement : Comparison of Marathon and Enduron polyethylene
- Total: Total of all reporting groups
Arm/Group | Crosslinked Marathon Polyethylene | Standard Enduron Polyethylene | Total
Number analyzed (Participants) | 116 | 114 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.6) | 62.0 (11.1) | 62.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 57 | 122
  Male | 51 | 57 | 108
Region of Enrollment [Number; unit: participants]
  United States | 116 | 114 | 230

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinically Significant Osteolysis
Description: The incidence of clinically significant osteolysis was based on the number of unrevised THAs (total hip arthroplasties) with at least 1.5 square centimeters of pelvic and/or femoral osteolysis. Osteolysis was defined as an area of localized loss of trabecular bone or cortical erosion that was not apparent on the pre-operative or immediate postoperative radiograph. To obtain lesion sizes, the defects were outlined on the anteroposterior pelvic radiograph and the area of the lesion was measured using Martell's Hip Analysis Suite software. Lesions were considered clinically important if the total area of osteolysis around a hip replacement was at least 1.5 square centimeters.
Time Frame: Minimum 9-year radiographic follow-up
Population: Minimum 9-year radiographs used to assess osteolysis were available for 79 unrevised hips with Marathon and 68 unrevised hips with Enduron polyethylene.
Measure: Number; unit: unrevised THAs
Arm/Group | Crosslinked Marathon Polyethylene | Standard Enduron Polyethylene
Number analyzed (Participants) | 79 | 68
unrevised THAs | 0 | 15

2. Secondary Outcome: Polyethylene Wear
Description: A single reviewer, who was blinded to the type of polyethylene liner, evaluated femoral head penetration among all unrevised hips with minimum 9-year radiographic follow-up using serial anteroposterior pelvic radiographs. Two-dimensional head penetration was determined for each follow-up radiograph relative to the immediate post-operative (nominal 6-week follow-up) reference view using Hip Suite Analysis version 8.0 with elliptical correction, a validated, computer-assisted technique. A linear wear rate was evaluated for each hip that had a minimum of three follow-up radiographs by using a least-squares linear regression to calculate the slope of the best-fit line for the wear vector magnitude versus time in situ data. The slope from this regression represented the steady-state linear wear rate. The steady-state linear wear rate data from all hips in a group was used to compute a mean polyethylene wear value.
Time Frame: Minimum 9-year radiographic follow-up
Population: At least 3 head penetration measurements evaluated with Martell's Hip Suite Analysis software were available for 76 unrevised hips with Marathon and 66 unrevised hips with Enduron polyethylene.
Measure: Mean (Standard Deviation); unit: millimeters per year
Arm/Group | Crosslinked Marathon Polyethylene | Standard Enduron Polyethylene
Number analyzed (Participants) | 76 | 66
millimeters per year | .04 (.06) | 0.22 (0.13)

3. Secondary Outcome: Rate of Reoperation
Description: The rate of reoperation was based on the number of reoperations in each group. Any additional surgery after a participant's initial hip replacement was considered a reoperation.
Time Frame: 10-year follow-up
Population: All 116 hips randomized to Marathon polyethylene and all 114 hips randomized to Enduron polyethylene were included in the analysis population to determine the rate of reoperation.
Measure: Number; unit: THAs
Arm/Group | Crosslinked Marathon Polyethylene | Standard Enduron Polyethylene
Number analyzed (Participants) | 116 | 114
THAs | 2 | 11

4. Secondary Outcome: Harris Hip Score
Description: The Harris Hip Score measures outcome after hip replacement and is based on a scale from 0 (worst) to 100 (best).
Time Frame: Minimum 9-year follow-up
Population: Harris Hip Scores were evaluated for 74 unrevised hips with Marathon and 65 unrevised hips with Enduron polyethylene that had minimum 9-year follow-up and complete data to compute a score.
Measure: Mean (Standard Deviation); unit: score on a 100 point scale
Arm/Group | Crosslinked Marathon Polyethylene | Standard Enduron Polyethylene
Number analyzed (Participants) | 74 | 65
score on a 100 point scale | 88 (14) | 86 (15)

5. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction was quantified by asking participants to respond "yes" or "no" to the question, "Are you satisfied with the results of your hip operation?"
Time Frame: Minimum 9-year follow-up
Population: Satisfaction rates were evaluated among 84 participants with unrevised hips who had Marathon and 70 participants with unrevised hips who had Enduron polyethylene. These participants had minimum 9-year follow-up and responded to the question about satisfaction.
Measure: Number; unit: percentage of participants
Groups:
- Crosslinked Marathon Polyethylene: Implanted with a metal femoral head and crosslinked polyethylene liner.
Arm/Group | Crosslinked Marathon Polyethylene | Standard Enduron Polyethylene
Number analyzed (Participants) | 84 | 70
percentage of participants | 99 | 97

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the duration of the study. The mean follow-up for the participants who were not revised and did not pass away within 9 years of their hip replacement was 10 years.
Description: Serious adverse events were collected by questioning study participants and reviewing medical records. The denominator for "Other (non-serious) Adverse Events" is listed as 0 because other (non-serious) Adverse Events were not collected/assessed.
Arm/Group | Crosslinked Marathon Polyethylene | Standard Enduron Polyethylene
Serious Adverse Events (participants affected / at risk) | 2/116 | 11/114
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crosslinked Marathon Polyethylene (N=116) | Standard Enduron Polyethylene (N=114)
Dislocation and Reoperation (Musculoskeletal and connective tissue disorders) | 2 | 2
Revision due to Wear/Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor requires at least 30 days to review and comment on manuscripts before submission. For abstracts, the time frame for review is at least 10 days before submission. The sponsor will inform the investigator of any changes deemed necessary to preserve the confidentiality of proprietary information or to ensure scientific accuracy.